CLINICAL TRIAL: NCT01066000
Title: A Single Arm Open Label Interventional Study to Assess the Efficacy, Safety and Tolerability of Once-monthly Administration of Intravenous Methoxy-polyethylene Glycol-epoetin Beta for the Maintenance of Haemoglobin Levels in Dialysis Patients With Chronic Renal Anaemia
Brief Title: A Study for Monthly Methoxy Polyethylene Glycol-Epoetin Beta Treatment in Patients With Chronic Renal Anaemia
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML21736
Record Dates: First submitted 2010-02-09; First posted 2010-02-10 (Estimated); Results first posted 2016-05-13 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — continuous erythropoietin receptor activator

ARMS (1):
- Mircera (Experimental)
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta [Mircera]

INTERVENTIONS:
Drug: methoxy polyethylene glycol-epoetin beta [Mircera] — initial doses of either 120 micrograms or 200 micrograms or 360 micrograms, once monthly

SUMMARY:
This open-label single-arm study will evaluate the efficacy, safety and tolerability of methoxy polyethylene glycol epoetin beta on long-term maintenance of haemoglobin levels in patients with chronic renal anaemia. Patients will receive methoxy polyethylene glycol-epoetin beta intravenously once monthly at initial doses of either 120 micrograms or 200 micrograms or 360 micrograms in the titration phase of 16 weeks with a potential dose adjustment in the evaluation phase of 8 weeks. The anticipated time on study treatment is 24 weeks. The target sample size is 50-100 patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults >/=18 years of age
* Chronic renal anaemia
* Haemoglobin concentration between 10 and 12 g/dL at screening
* Adequate iron status
* Continuous intravenous maintenance short-acting therapy with same dosing interval for 8 weeks prior to screening
* Regular long-term haemodialysis therapy for at least 12 weeks prior to screening

Exclusion Criteria:

* Change in haemoglobin concentration >/=2 g/dL during screening
* Transfusion of red blood cells less than 8 weeks prior to screening
* Poorly controlled hypertension
* Relevant acute or chronic bleeding requiring treatment less than 8 weeks prior to screening
* Active malignant disease
* Haemolysis
* Haemoglobinopathies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2009-10-31 (Actual); Primary Completion 2011-09-30 (Actual); Study Completion 2011-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (12):
- Indonesia (12):
  - Advent Hospital; Kidney and Hipertension, Bandung
  - Sanglah Hospital; Kidney and Hipertension, Denpasar
  - Rumah Sakit Pgi Cikini; Renal & Hypertension, Jakarta
  - Cipto Mangunkusumo Hospital; Renal and Hypertension division, Internal Medecine Department, Jakarta
  - Pelni Hospital; Kidney and Hipertension, Jakarta
  - Pondok Indah Hospital; Kidney and Hipertension, Jakarta
  - Pantai Indah Kapuk Hospital; Kidney and Hipertension, Jakarta
  - Klinik Spesialis Ginjal dan hipertensi Rasyida; Renal and Hypertension, Medan
  - Pirngadi; Renal and Hypertension, Medan
  - Telogorejo Hospital; Renal and Hypertension, Semarang
  - Dokter Soetomo Hospital, Surabaya
  - PHC Hospital; Renal and Hypertension, Surabaya

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 10 sites in the Indonesia and the study period was from 05 October 2009 to 12 September 2011.
Pre-assignment Details: Of the 85 screened participants 52 were screening failure due to abnormal haemoglobin concentration and 33 were enrolled in the study.
Groups:
- Mircera: Eligible participants received methoxy polyethylene glycol-epoetin beta (Mircera) intravenously (IV), once every four weeks for 24 weeks. Participants received a starting dose of Mircera 100, 150 or 200 microgram (mcg) which was based on the Epoetin dose of<8000, 8000-16000, or >16000 International units [IU]/Week, administered during the week preceding the switch to the study drug.
Period: Overall Study
Arm/Group | Mircera
Started | 33
Completed | 24
Not Completed | 9
Not completed — Protocol Violation | 4
Not completed — Death | 3
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- Mircera: Eligible participants received Mircera IV, once every four weeks for 24 weeks. Participants received a starting dose of Mircera 100, 150 or 200 mcg which was based on the Epoetin dose of <8000, 8000-16000, or >16000 IU/Week, administered during the week preceding the switch to the study drug.
Arm/Group | Mircera
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.7 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 20

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Maintaining Average Haemoglobin During the Efficacy Evaluation Period Within the Target Range (10-12 g/dl)
Description: The proportion of participants with their mean haemoglobin (Hb) concentration (g/dL) within the target range during the efficacy evaluation period was assessed. The target range is the reference Hb not >12 g/dL and not < 10 g/dL.
Time Frame: Up to Week 24
Population: Intent to treat (ITT) population was defined as all participants who entered study and took at least one dose of study drug. The ITT and safety population were identical. At Week 24, data of 24 participants were included whereas 9 participants were excluded from the analysis as they discontinued the study before analysis of this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Mircera
Number analyzed (Participants) | 24
Percentage of participants | 45.8

2. Secondary Outcome: Number of Participants With Adverse Events and Serious Adverse Events
Description: An adverse event (AE) was defined as any untoward medical occurrence that occurred during the course of the trial after study treatment had started. An adverse event was therefore any unfavourable and unintended sign, symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug. A Serious adverse event (SAE) is any untoward medical occurrence that at any dose results in death, are life threatening, requires hospitalization or prolongation of hospitalization or results in disability/incapacity, and congenital anomaly/birth defect. The AEs were assessed from baseline to every visit throughout the treatment, post study drug discontinuation, and follow up period.
Time Frame: Up to Week 28
Population: Safety population included all participants who entered into the study and took at least one dose of study drug.The ITT and safety population were identical. Data of maximum number of participants (33 participants) available at the time of analysis were analysed and reported.
Measure: Number; unit: Participants
Arm/Group | Mircera
Number analyzed (Participants) | 33
Participants
  Number of participants serious AE | 4
  Total number of participants with at least one AE | 15

3. Secondary Outcome: Mean Change in Haemoglobin Concentration From Screening Period and Efficacy Evaluation Period
Description: The mean haemoglobin (Hb) concentration (g/dL) change from the baseline (Week 0) till efficacy evaluation period (EEP) was assessed and reported.
Time Frame: Up to Week 24
Population: ITT population was defined as all participants who entered study and took at least one dose of study drug. The ITT and safety population were identical. At Week 24, data of 24 participants were included whereas 9 participants were excluded from the analysis as they discontinued the study before analysis of this outcome measure.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Mircera
Number analyzed (Participants) | 24
g/dL
  At baseline | 10.89 (0.48)
  Mean change at EEP | 0.04 (1.23)

4. Secondary Outcome: Proportion of Participants Maintaining Haemoglobin Concentration Within the Haemoglobin Range 10-12g/dL Throughout the Efficacy Evaluation Period
Description: The proportion of participants maintaining haemoglobin concentration within the haemoglobin range 10-12g/dL throughout the efficacy evaluation period (EEP) was assessed and reported.
Time Frame: Up to Week 24
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Mircera
Number analyzed (Participants) | 24
Percentage of participants
  Participants maintaining Hb >10 g/dl | 62.5
  Participants maintaining Hb within 10-12 g/dl | 16.7

5. Secondary Outcome: Mean Time Spent by Participants in the Haemoglobin Range of 10 - 12 g/dL During the Efficacy Evaluation Period
Description: Mean time spent in the haemoglobin range 10 - 12 g/dL during the efficacy evaluation period (EEP) was assessed and reported.
Time Frame: Up to Week 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Mircera
Number analyzed (Participants) | 24
Weeks | 3.92 (2.39)

6. Secondary Outcome: Mean Number of Months Per Participant Requiring Dose Adjustment During the Dose Titration and Evaluation Periods
Description: Mean number of months per participant requiring dose adjustment during the dose titration and evaluation periods was assessed and reported.
Time Frame: Up to Week 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Mircera
Number analyzed (Participants) | 24
Months | 1 (3.5)

7. Secondary Outcome: Mean Monthly Dose of Methoxy Polyethylene Glycol-epoetin Beta During the Dose Titration and Evaluation Periods
Description: Mean monthly dose of methoxy polyethylene glycol-epoetin beta during the dose titration and evaluation periods was assessed and reported.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 16, and Week 20
Population: ITT population was defined as all participants who entered into study and took at least one dose of study drug. The ITT and safety population were identical. Data of maximum number of participants (24 participants) available at the time of analysis were analysed and 9 participants discontinued the study before this analysis.
Measure: Mean (Standard Deviation); unit: μg/month
Arm/Group | Mircera
Number analyzed (Participants) | 24
μg/month
  At Baseline | 97.9 (14.6)
  At Week 4 | 103.1 (19.9)
  At Week 8 | 107.3 (37.9)
  At Week 12 | 119 (43.8)
  At Week 16 | 114.6 (53.6)
  At Week 20 | 120.8 (73.2)

8. Secondary Outcome: Number of Participants With Marked Laboratory Abnormalities
Description: A marked laboratory abnormality is defined as above and/or below the normal range of a laboratory parameter which was considered to be potentially clinically relevant. The number of participants with marked laboratory abnormality are presented. Marked laboratory abnormalities were analyzed according to the Roche specified limits for the following reference range: Haemoglobin (Hb) (11.7-17.3 g/dL), Haematocrit (Hct) (35-47%), White blood cells (WBC) (3.6-11.0 10^3/µL), Red blood cells (RBC) (3.8- 5.9 10^6/µL), MCV (80-100 fL) Platelets (150-440 10^3/µL), Iron (37-158 µg/dL), Ferritin (10-365 ng/mL), Transferrin (170-340 mg/dL), TIBC (250-450 µg/dL), TSAT (15-50%), Albumin (3.4-4.8 g/dL), hs-CRP (<= 10.000 mg/dL), Potassium (3.5-5.1 mmol/L), and Phosphorus (2.7-4.5 mg/dL).
Time Frame: Up to Week 28
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Mircera
Number analyzed (Participants) | 33
Participants
  At Baseline, Hb-Low | 30
  At Baseline, Hct-Low | 28
  At Baseline, WBC-Low | 1
  At Baseline, WBC-High | 2
  At Baseline, MCV-Low | 3
  At Baseline, MCV- High | 4
  At Baseline, RBC-Low | 1
  At Baseline, RBC -High | 2
  At Baseline, Platelets-Low | 7
  At Baseline, Iron-Low | 10
  At Baseline, Iron-High | 1
  At Baseline, Feritin-High | 25
  At Baseline, Transferin-Low | 9
  At Baseline, TIBC-Low | 24
  At Baseline, TSAT-Low | 8
  At Baseline, TSAT-High | 8
  At Baseline, Albumin-Low | 3
  At Baseline, hs-CRP-High | 2
  At Baseline, Potassium-High | 9
  At Baseline, Phosphorus-High | 19
  At Week 8, Hb-Low | 22
  At Week 8, Hct-Low | 22
  At Week 8, WBC-High | 3
  At Week 8, MCV-Low | 5
  At Week 8, RBC -High | 25
  At Week 8, Platelets-Low | 1
  At Week 8, Platelets-High | 21
  At Week 8, Iron-Low | 1
  At Week 8, Iron-High | 22
  At Week 8, Feritin-High | 6
  At Week 8, Transferin-Low | 6
  At Week 8, TIBC-Low | 24
  At Week 24, Hb-Low | 18
  At Week 24, Hct-Low | 14
  At Week 24, WBC-High | 2
  At Week 24, RBC -High | 4
  At Week 24, Platelets-Low | 4
  At Week 24, Platelets-High | 1
  At Week 24, Iron-Low | 4
  At Week 24, Iron-High | 1
  At Week 24, Feritin-High | 8
  At Week 24, Transferin-Low | 6
  At Week 24, Transferin-High | 1
  At Week 24, TIBC-Low | 12
  At Week 24, TSAT-Low | 1
  At Week 24, TSAT-High | 3
  At Week 24, Albumin-High | 1
  At Week 24, hs-CRP-High | 2
  At Week 24,Potassium-Low | 2
  At Week 24, Potassium-High | 3
  At Week 24, Phosphorus-High | 11

ADVERSE EVENTS:
Time Frame: Up to 28 weeks
Description: Serious adverse events and non-serious adverse events are reported in Safety Analysis Set, which consists of all participants who received at least one dose of study medication and had a safety assessment performed post baseline.
Arm/Group | Mircera
Serious Adverse Events (participants affected / at risk) | 4/33
Other Adverse Events (participants affected / at risk) | 15/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mircera (N=33)
Decrease of state awareness (Nervous system disorders) | 1
Colic renal (Renal and urinary disorders) | 1
Cardiovascular event (Cardiac disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mircera (N=33)
Hepatitis (Infections and infestations) | 1
Fever (General disorders) | 1
Headache (Nervous system disorders) | 3
Dizziness (Nervous system disorders) | 1
Decrease of state of awareness (Nervous system disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Haemorrhoid (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Itching (Skin and subcutaneous tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Allergy (Immune system disorders) | 1
Food allergy (Immune system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Cardiovascular event (Cardiac disorders) | 1
Menstruate (Reproductive system and breast disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Hematuria (Renal and urinary disorders) | 2
Colic renal (Renal and urinary disorders) | 1

LIMITATIONS AND CAVEATS:
This was an open-label, single arm study with no control arms for comparison of results from this study.

The study was prematurely terminated due to high screening failures and low recruitment rate. Therefore, the data only showed a trend.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.